CLINICAL TRIAL: NCT06690788
Title: PreventT2 Together: Examining the Efficacy of Couple-based Lifestyle Intervention to Prevent Type 2 Diabetes
Acronym: PT2T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katherine Baucom, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 166946; 1R01DK140177-01 (NIH)
Record Dates: First submitted 2024-08-12; First posted 2024-11-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prediabetic State; Life Style; Intervention Study; Social Support; Physical Activity; Obesity
Keywords: Lifestyle Intervention; Prevention; Social Support; Couple Relationships
MeSH Terms: conditions — Prediabetic State; Motor Activity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual intervention condition (Active Comparator): "PreventT2" individual lifestyle intervention curriculum (2021 revised National DPP curriculum, freely available from the CDC)
  Interventions: Behavioral: Individual intervention condition (PreventT2)
- Couple-based intervention condition (Experimental): "PreventT2 Together" (couple-based adaptation of PreventT2; approved by the CDC in November 2022 as an Alternate Curriculum for use in the National DPP)
  Interventions: Behavioral: Couple-based intervention condition (PreventT2 Together; couple-based adaptation of 2021 PreventT2; approved by the CDC in November 2022 as an Alternate Curriculum for use in the NDPP)

INTERVENTIONS:
Behavioral: Individual intervention condition (PreventT2) — PreventT2 will be delivered by a team of trained CDC National Diabetes Prevention Program (NDPP) Lifestyle Coaches to adults at high risk for diabetes. The 2021 version of the lifestyle intervention curriculum to be used is freely available from the CDC. The intervention will be delivered in the context of the University of Utah National DPP, which has Full recognition from the CDC based on outcome data over the course of a number of years.
  Arms: Individual intervention condition
Behavioral: Couple-based intervention condition (PreventT2 Together; couple-based adaptation of 2021 PreventT2; approved by the CDC in November 2022 as an Alternate Curriculum for use in the NDPP) — PreventT2 Together will be delivered by a team of trained CDC National DPP Lifestyle Coaches to adults at high risk for diabetes and their partners. The lifestyle intervention curriculum was developed with the input of a community advisory board and was approved by the CDC for use in the National DPP (Diabetes Prevention Program) (i.e., meets CDC Diabetes Prevention Recognition Program Standards, including 22+ classes delivered over the course of 12 months and targeting lifestyle changes to prevent type 2 diabetes). In contrast to PreventT2, the intervention includes content specific to couples with prompts encouraging partners to consider and discuss how they can best support one another, information about lifestyle intervention in a relationship context, and examples demonstrating how couples collaborated to make healthy lifestyle changes.
  Arms: Couple-based intervention condition

SUMMARY:
Nearly half of adults in the United States have or are at risk of developing type 2 diabetes. The overall goal of this community-engaged research is to examine the efficacy of an innovative couple-based lifestyle intervention to prevent type 2 diabetes that is applicable to a broad range of partnered adults in the United States. By simultaneously targeting lifestyle and perceived support from romantic partners, there is a high likelihood of creating lasting changes in both

DETAILED DESCRIPTION:
Nearly half of U.S. adults have or are at risk of developing type 2 diabetes. Lifestyle intervention is efficacious and the first line of prevention among adults at high risk for type 2 diabetes. Unfortunately, outcomes in real-world settings do not approach the initial efficacy trial findings, in part due to low rates of retention in the intervention. Real-world programs have particularly struggled to retain participants who identify as members of racial/ethnic groups that are disproportionately affected by type 2 diabetes, potentially exacerbating health disparities. Given the strong influence romantic partners have on one another and the shared environment, in which couples typically live, lifestyle interventions that systematically include romantic partners have the potential to address the research-practice gap. The purpose of this project is to examine the efficacy of PreventT2 Together, a couple-based lifestyle intervention our team developed. The specific aims of the research are: (1) to determine the efficacy of PreventT2 Together in a single-center, randomized clinical trial,(2) to examine baseline relationship satisfaction as a moderator and perceived partner support as a mechanism of lifestyle change, and (3) to quantify intervention retention and describe reach across recruitment methods. The investigators will recruit 162 couples (i.e., adults at high risk for type 2 diabetes and their romantic partners)from community and healthcare settings, over-sampling members of racial/ethnic minority groups. The investigators will randomize participating couples to individual (PreventT2; delivered only to partners at high risk) or couple-based (PreventT2 Together; delivered to couples) lifestyle intervention conditions. HbA1c and objectively measured moderate to vigorous physical activity (MVPA) will be collected from all participants at baseline (Pre)and at the end of the 1-year intervention (Post). Participants will also report on lifestyle factors, health outcomes, and relationship functioning at each of 13-time points (Pre, monthly, during the intervention, and post). The investigators focus on the patient-centered minimum clinically important difference (MCID) in outcomes, including objectively-measured MVPA (primary outcome), as well as other aspects of lifestyle (nutrition, sleep), health outcomes (HbA1c, weight loss, stress), and relationship functioning (perceived partner support) (secondary outcomes). Situating lifestyle intervention within the romantic relationship context in which lifestyle change occurs is likely to increase reach and improve retention and lifestyle change outcomes in real-world settings. Our community-engaged approach to the development of the intervention and design of the proposed project will ensure broad applicability and dissemination of results across communities, including racial/ethnic minority groups that have not been effectively reached and retained. CDC review and approval of PreventT2 Together for use as an alternate curriculum in the National Diabetes Prevention Program (National DPP) delivered across the U.S. underscores the scalability of the intervention. If efficacious, PreventT2 Together has the potential to impact individuals and their romantic partners' quality of life and ultimately improve real-world outcomes of lifestyle intervention to prevent type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. "Target partner" is eligible for the National DPP per CDC eligibility requirements:

   * BMI ≥ 25 kg/m² (≥ 23 kg/m² if Asian American), and
   * Do not have a diagnosis of type 1 or type 2 diabetes, and
   * Not currently pregnant, and
   * High risk for type 2 diabetes based on: (i) CDC Prediabetes Risk Test score ≥ 5, (ii) clinically diagnosed Gestational Diabetes during a previous pregnancy (for women), or (iii) a blood test result indicative of prediabetes in the past year (i.e., fasting blood glucose 100-125 mg/dl; plasma glucose 140-199 mg/dl measured 2 hours after a 75 g glucose load; or HbA1c 5.7%-6.4%).
2. The couple has lived together for 1+ years.
3. Both partners are willing to participate in the research.
4. Both partners are at least 18 years old.
5. Both partners are fluent in English.

EXCLUSION CRITERIA:

1. "Supporting partner" has a diagnosis of Type 2 Diabetes.
2. Either partner:

   * Has a diagnosis of another chronic disease (unless no major events/changes for 3+ months), or
   * Is currently on medication or engaged in lifestyle intervention for prediabetes or obesity, or
   * Has previously participated in the National DPP, or
   * Reports discomfort participating in a lifestyle program with their partner, or
   * Reports a low level of relationship commitment (i.e., "4" or lower on a scale from 1 (do not agree at all) to 7 (agree completely) on the item "I want this relationship to stay strong no matter what rough times we encounter."; Owen et al., 2011).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Percent of target partners achieving clinically meaningful increases in Moderate to Vigorous Physical Activity (MVPA) | 14 months
  International Physical Activity Questionnaire (IPAQ)-7 day (Pre-Intervention, Post-Intervention) and a 7-day At-Home accelerometer assessment (Pre-Intervention, Post-Intervention). International Physical Activity Questionnaire (IPAQ)-7 day (Monthly during Intervention). Among participants attending intervention classes, starting at the fourth class minutes of moderate-to-vigorous physical activity (MVPA) over the past week will be reported to Lifestyle Coaches. International Physical Activity Questionnaire (IPAQ) questionnaires assess self-reported walking, moderate intensity, and vigorous intensity physical activity as well as overall sedentary time. Accelerometers provide objective assessments of these constructs. Intervention class participants self-report the total number of Moderate to Vigorous Physical Activity (MVPA) minutes over the previous week.

SECONDARY OUTCOMES:
HbA1c | 14 months
  Assessed by the research team using the A1c Now Point of Care System.
Weight | 14 months
  Weight in pounds will be assessed by the research team at both the Pre and Post time points using a medical grade scale. Among participants attending intervention classes, weight in pounds will be privately measured by Lifestyle Coaches before each class.
Stress | 14 months
  Assessed with the Perceived Stress Scale measure (Possible score range: 0-24, with higher scores representing higher levels of perceived stress).
Nutrition | 14 months
  Assessed with the Automated self-administered 24-hr recall (ASA24) (Pre, Post). We will examine the following outcomes: Healthy Eating Index (HEI), total vegetable, added sugars, fiber, whole grains, refined grains, and total KiloCalorie. (HEI Score Range: 0-100, with higher scores representing sets of foods that more closely align with key dietary recommendations and patterns.)(Total Vegetable expressed in cups, added sugars expressed in teaspoon equivalents, fiber expressed in grams, whole grains expressed in ounce equivalents, refined grains expressed in ounce equivalents, and total KCal expressed in kilocalories.)
  Assessed with the Rapid Eating and Activity Assessment for Participants (REAP-S; Composite Score Range 13-39, with higher scores representing higher diet quality) (Monthly).
Sleep | 14 months
  Assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Version 1.0 Sleep-Related Impairment 8a (T-score range: 30-80.1, with higher scores indicating higher levels of sleep-related impairment) and the PROMIS Short Form Version 1.0 Sleep Disturbance 8a (T-score range: 30.5-77.5, with higher scores indicating higher levels of sleep disturbance).
Perceived Partner Support | 14 months
  Assessed with the Multidimensional Scale of Perceived Social Support "special person" subscale, with the language updated to "romantic partners," consistent with prior work. This subscale assesses the amount of support individuals perceive from their romantic partners (Score range: 4-28, with higher scores indicating more perceived support from romantic partners).

OTHER OUTCOMES:
Anxiety | 14 months
  Assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Version 1.0 Anxiety 8a (T-score range: 37.1-83.1, with higher scores indicating higher levels of anxiety symptoms).
Depression | 14 months
  Assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Version 1.0 Depression 8a (T-score range: 38.2-81.3, with higher scores indicating higher levels of depressive symptoms).
Fatigue | 14 months
  Assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Fatigue 7a (T-score range: 29.4-83.2, with higher scores indicating higher levels of fatigue).
Relationship Satisfaction | 14 months
  Assessed with the Couples Satisfaction Index-16 (CSI-16), a measure of overall relationship satisfaction (Score range: 0-81, with higher scores indicating higher levels of relationship satisfaction).
Interest in Sexual Activity | 14 months
  Assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale Version 2.0 Sexual Function and Satisfaction: Interest in Sexual Activity (T-score range: 21.9-65.8, with higher scores indicating more interest in sexual activity).
Intervention Attendance | 12 months
  Lifestyle Coaches will record whether participants attend each intervention class. Total intervention attendance will be the total number of classes attended in-person (make-up classes, while offered to participants who miss the in-person class, will not count toward this total).
Lifestyle Coach Fidelity | 12 months
  A DTTAC Master Trainer Select will rate Lifestyle Coach fidelity in 10% of classes.
Additional lifestyle intervention engagement | 12 months
  Participants will respond to a single item on the questionnaire regarding whether they received additional lifestyle intervention to supplement National DPP classes. If yes, they will be asked to describe what they did as well as the frequency and duration of the intervention.
Intervention Retention | 12 months
  Intervention Retention will be measured by whether participants meet CDC criteria for "completer" status (i.e., attend at least 9 total classes, with at least 8 classes in the first six months of the program, and at least 1 class in the second six months of the program that occurs 9 months following the first class).
Percent of individuals approached who are eligible and enroll in the study (Reach) | 14 months
  Reach will be measured by (a) the percent of individuals approached who are eligible and enroll in the study.
Intervention Acceptability | 14 months
  Acceptability of the individual and couple-based lifestyle interventions will be measured with the Theoretical Framework of Acceptability-Based Questionnaire
Pain Interference | 14 months
  Assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Short Form Version 1.0 4a (T-score range: 41.6 - 75.6 with a higher score indicating more pain interference.)
Daily Report of Social Control | 14 months
  Assessed with the Daily Report of Social Control Measure (Score Range 1-2 with lower scores indicating more Social support from partners.)
Communal Coping | 14 months
  Assessed with the Theoretical Model of Communal Coping (TMCC) Appraisal and Action Subscales. (Score Range of 33-50, with higher scores indicating more shared appraisal or action.)
The Accountable Health Communities Screening Tool | 14 months
  Assessed with the Accountable Health Communities Core Health-Related Social Needs Screening Questions. (No score range, but underlined answer options indicate positive responses for the associated health-related social need.)
Health Care Access and Preventive Health Screenings | 14 months
  Assessed with questions from the National Health Interview Survey (NHIS.) (No Score Range, but questions indicate health care access, occurrence of preventive health screenings, as well as delay or missing health care intervention due to cost avoidance.)
Percent of supporting partners who enroll in the study that are at high risk for type 2 diabetes based on the Pre HbA1c and self-report questionnaires (Reach) | 14 months
  Reach will be measures by the percent of supporting partners who enroll in the study that are at high risk for type 2 diabetes based on the Pre HbA1c and self-report questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Katherine JW Baucom, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguirre MC, Brown H, Gershenoff D, Hinton KL, Huntzinger OM, Klein N, Ramos C, Tavake-Pasi OF, Witte B, Wolfsfeld M, Sher T, Simmons DL, Smith TW, Clark L, Baucom KJW. The Role of Advocacy in Adapting the Diabetes Prevention Program for Couple-Based Delivery That Reaches Marginalized Groups. Behav Ther (N Y N Y). 2020 Oct;43(7):261-265. No abstract available. PMID 33536698
- [Background] Whitaker M, Aguirre MC, Gutierrez Chavez M, Beaulieu E, Arones YB, Gershenoff D, Hinton K, Klein N, Munezerou Uwizeye J, Napia E, Ramos C, Tavake-Pasi OF, Villalta J, Wolfsfeld C, Witte B, Maxfield E, Raphael K, Simmons DL, Clark L, Sher T, Smith TW, Baucom KJ. Couple-based lifestyle intervention to prevent type 2 diabetes: protocol for a randomised pilot trial. BMJ Open. 2023 Feb 16;13(2):e068623. doi: 10.1136/bmjopen-2022-068623. PMID 36797025